CLINICAL TRIAL: NCT02313025
Title: Spreken Verfijnen in de Kleuterklas: De Ontwikkeling Van Een Spraakdidactiek Als Uitbreiding op de Gangbare Taaldidactiek in Het Kleuteronderwijs
Brief Title: A Speech Sound and Phonemic Awareness Intervention in Flemish Early Childhood Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Lieve Van Severen, dr., KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CatholicULeuven
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Other Developmental Disorders of Speech and Language
MeSH Terms: conditions — Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Speech sound intervention (Experimental): This group receives a speech sound and phonemic awareness intervention for four months.
  Interventions: Other: speech sound intervention
- World-project (Active Comparator): This group receives the WORLD intervention for four months.
  Interventions: Other: World-project

INTERVENTIONS:
Other: speech sound intervention — An intervention that stimulates speech sound perception and production in four-year-olds.
  Each day at preschool the children receive a 15 to 20 minutes intervention, for 12 weeks
  Other Names: Kaatje Klank
  Arms: Speech sound intervention
Other: World-project — An intervention that stimulates vocabulary development in four-year-olds. Each day at preschool the children receive a 120 minutes intervention, for 10 weeks
  Other Names: Wereldwoorden
  Arms: World-project

SUMMARY:
The language intervention 'Kaatje Klank' is designed for stimulating the speech production and speech perception skills of 4-year-olds in an early childhood educational setting, in order to stimulate early literacy skills. These skills are crucial skills for technical reading in later ages. Good reading skills are an important condition for academic success.

To measure the effect of the language intervention 'Kaatje Klank', the intervention will be applied in six Dutch preschool classes (n = 100 children, 50% native speakers of Dutch, 50% non-native speakers) during 12 weeks (daily). Teachers will be trained and observed using a coaching trajectory.To measure the effect on speech production and perception skills, a pre- and posttest and a comparison with a matched control group (n = 100 children, 50% native speakers of Dutch, 50% non-native speakers) will be used. The control group will receive a different language intervention which focuses on vocabulary development (World-project).

ELIGIBILITY:
Inclusion Criteria:

* In eary childhood education in Flanders (2de kleuterklas)

Exclusion Criteria:

* Language or speech disorder
* Less than 1 year acquiring Dutch

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
test battery: speech articulation test + phonemic awareness | Participants will be tested after an intervention of 12 weeks. The expected average test duration is 16 minutes

SECONDARY OUTCOMES:
vocabulary test (Wereldwoorden project) | Participants will be tested after an intervention of 12 weeks. The expected average test duration is 4 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lieve Van Severen, Dr, Principal Investigator — KU Leuven
Locations (1):
- Odisee, Aalst, Oost-Vlaanderen, Belgium

REFERENCES:
- See also: Information on the speech sound intervention — http://www.kaatjeklank.be